CLINICAL TRIAL: NCT02729909
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lubiprostone for the Treatment of Chronic Idiopathic Constipation
Brief Title: Lubiprostone for Chronic Idiopathic Constipation Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lubiprostone-3003; U1111-1168-6358 (Registry Identifier: WHO); 153300410A0196 (Registry Identifier: RNEC)
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Constipation
Keywords: Drug therapy
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lubiprostone 24 μg (Experimental): Lubiprostone 24 μg, capsules, orally, twice daily, under fed conditions, for 4 weeks.
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Lubiprostone placebo-matching capsules, orally, twice daily, under fed conditions, for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone capsules
  Other Names: AMITIZA
  Arms: Lubiprostone 24 μg
Drug: Placebo — Lubiprostone placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of oral administration of 24 ug of lubiprostone twice daily (BID) for 4 weeks in participants with chronic idiopathic constipation (CIC) compared with placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called lubiprostone. Lubiprostone is being tested to treat people who have chronic idiopathic constipation. This study will look at the frequency of spontaneous bowel movements (SBMs) in people who take lubiprostone compared to placebo.

The study will enroll approximately 211 participants. Participants will be randomly assigned (by chance, like flipping a coin) equally to one of the two treatment groups, which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Lubiprostone 24 μg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

All participants will be asked to take one capsule with breakfast and one capsule with dinner each day throughout the study. All participants will be asked to record each time they have a SBM and all details of each SBM (including the consistency of the stool and the difficulty they have in passing it) in a diary.

This multi-center trial will be conducted in Mexico. The overall time to participate in this study is 8 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a history of constipation defined as having spontaneous bowel movement (SBM) frequency of less than 3 times per week on average for 6 months or longer and for whom the same SBM frequency is observed during the Screening Period.
4. Has had 1 or more of the symptoms associated with SBM (described below) for 6months or longer at the start of Screening:

   1. Scybalum stool or hard feces in at least 1 out of every 4 bowel movements.
   2. Sensation of incomplete evacuation in at least 1 out of every 4 bowel movements.
   3. Straining in at least 1 out of every 4 bowel movements.
5. Rarely has loose stools without the use of laxatives.
6. Is willing and able to keep a diary on his/her own and willing and able to complete a questionnaire.
7. Is male or female and aged 18 years or older, at the time of signing an informed consent.
8. A female participant of childbearing potential who is sexually active agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and 14 days after the last dose of study drug.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received lubiprostone in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening.
5. Has a history or clinical manifestations of significant mechanical obstruction (intestinal obstruction due to tumor, hernia etc).
6. Has a history of hypersensitivity or allergies to lubiprostone or any of its excipients.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit.
8. Is required to take excluded medications.
9. If female, is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
10. Participant whose constipation is considered to be due to drugs or to whom a prohibited concomitant medication has been administered.
11. Is having chronic constipation due to a secondary cause (medications, diabetes mellitus, hypothyroidism, depression, etc.)
12. Has sufficient criteria for irritable bowel syndrome (IBS) or functional defecation disorder.
13. SBM frequency is 3 or more per week.
14. SBM frequency has been less than 3 times per week for less than 6 months in duration or whose symptoms associated with SBM have been present for less than 6 months (hard feces, sensation of incomplete evacuation, or straining).
15. Has received treatment with a rescue medication within 24 hours prior to the first dose on the morning of Day1: bisacodyl suppository, which is a standard laxative, glycerin enema, or any other rescue medication.
16. Has megacolon/megarectum or has received a diagnosis of intestinal pseudo-obstruction.
17. Has confirmed or suspected organic disorders of the large intestine (obstruction, stenosis, carcinoma, or inflammatory bowel disease). Organic disorders of the large intestine can be confirmed or ruled out using the results of enema X-ray examination or total colonoscopy performed in the previous 2 years. If the participant has no history or shows no current evidence of weight loss, anemia, or rectal bleeding, organic disorders may be ruled out based on the results of such testing performed in the past 3 years. Any participant in whom total colonoscopy has detected a polyp requiring treatment is excluded from this study .Note: Participant should not be screened unless at least 7 days have passed since an enema X-ray examination, total colonoscopy or sigmoidoscopy have been performed.
18. Has been hospitalized for gastrointestinal or abdominal surgery within 3 months prior to Screening.
19. Has a significant cardiovascular, liver, lung, kidney, neurological, or mental disease (including existing alcohol or drug abuse problem) or a systemic disease.
20. Has significant clinical findings or in whom a significant abnormality has been found in hematology test, serum chemistry, or urinalysis.
21. Participant in whom noncompliance with the study protocol (administration schedule, visit schedule, diary completion or other study procedure) is expected.
22. Has a history of malignant disease (except basal cell carcinoma) within 5 years prior to Screening.
23. Has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or total bilirubin >2.0 mg/dL with AST/ALT elevated above the limits of normal values.
24. Participant who the investigator/subinvestigator has determined ineligible to participate in this study for any reason other than the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- Mexico (10):
  - Mexicali, Baja California Norte
  - León, Guanajuato
  - Mexico City, Mexico City
  - Morelia, Michoacán
  - Monterrey, Nuevo Le0n
  - Culiacán, Sinaloa
  - Cuautitlán Izcalli, State of Mexico
  - Tlalnepantla, State of Mexico
  - Chihuahua City
  - Durango

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in Mexico from 11 May 2016 to 05 June 2017.
Pre-assignment Details: Participants with a diagnosis of chronic idiopathic constipation were enrolled in a 1:1 ratio in one of two treatment groups to receive either lubiprostone 24 µg or placebo.
Period: Overall Study
Arm/Group | Lubiprostone 24 μg | Placebo
Started | 105 | 106
Completed | 104 | 101
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Significant Protocol Deviation | 0 | 2
Not completed — Voluntary Withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total set included all participants who signed the informed consent form, including participants withdrawn prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone 24 μg | Placebo | Total
Number analyzed (Participants) | 105 | 106 | 211
Age, Continuous [Mean (Full Range); unit: years] | 43.3 [19 to 81] | 40.8 [18 to 84] | 42.05 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 90 | 172
  Male | 23 | 16 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 73 | 67 | 140
  White | 27 | 30 | 57
  Multiracial | 5 | 9 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 105 | 106 | 211
Height [Mean (Standard Deviation); unit: cm] | 161.9 (8.12) | 160.7 (7.42) | 161.3 (7.78)
Weight [Mean (Standard Deviation); unit: kg] | 72.48 (13.916) | 70.67 (12.873) | 71.57 (13.401)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.638 (4.6950) | 27.333 (4.3830) | 27.485 (4.5326)
Smokers [Count of Participants; unit: Participants]
  Participant had never smoked | 78 | 88 | 166
  Participant was a current smoker | 23 | 13 | 36
  Participant was an ex-smoker | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Bowel Movement (SBM) Frequency at Week 1 of Administration
Description: A SBM is defined as any bowel movement (BM) that does not occur within 24 hours after rescue medication use (laxative, suppository, or enema). Participants were given a diary to complete at home where they have recorded all details of each SBM including the consistency of the stool and the difficulty they have in passing it.
Time Frame: Week 1
Population: Full Analysis Set (FAS) included all participants randomized to receive study treatment whether or not they received treatment. Missing values were imputed by using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: number of SBM per week
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
number of SBM per week | 6.7 (4.55) | 5.2 (2.82)
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Test type: Superiority; p = 0.020, Van Elteren Test — Spontaneous bowel movement was analyzed using Van Elteren Test stratified by center. Centers with less participants were pooled based on geographical proximity; Median Value of confidence interval (CI) = 1.0, 95% CI 2-sided [0.1 to 1.9]

2. Secondary Outcome: SBM Frequency at Weeks 2, 3 and 4
Description: A SBM is defined as any BM that does not occur within 24 hours after rescue medication use (laxative, suppository, or enema). Participants were given a diary to complete at home where they have recorded all details of each SBM including the consistency of the stool and the difficulty they have in passing it.
Time Frame: Weeks 2, 3 and 4
Population: FAS included all participants randomized to receive study treatment whether or not they received treatment. Missing values were imputed by using LOCF.
Measure: Mean (Standard Deviation); unit: number of SBM per week
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
number of SBM per week
  Week 2 | 6.9 (4.40) | 5.5 (2.75)
  Week 3 | 7.6 (4.50) | 6.0 (3.74)
  Week 4 | 7.2 (4.21) | 5.8 (3.39)
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Week 2; Test type: Superiority; p = 0.051, Van Elteren Test — [p-value comment as in outcome 1, analysis 1]; Median Value of CI = 1.0, 95% CI 2-sided [0.0 to 1.9]
Statistical Analysis 2: Comparison: Lubiprostone 24 μg vs Placebo; Week 3; Test type: Superiority; p = 0.003, Van Elteren Test — [p-value comment as in outcome 1, analysis 1]; Median Value of CI = 1.5, 95% CI 2-sided [1.0 to 2.0]
Statistical Analysis 3: Comparison: Lubiprostone 24 μg vs Placebo; Week 4; Test type: Superiority; p = 0.009, Van Elteren Test — [p-value comment as in outcome 1, analysis 1]; Median Value of CI = 1.0, 95% CI 2-sided [0.1 to 1.9]

3. Secondary Outcome: Percentage of Participants Who Have a SBM Within 24 Hours After First Dose of Study Medication
Description: A SBM is defined as any BM that does not occur within 24 hours after rescue medication use. Percentage of participants who have an SBM within 24 hours after the first dose was assessed and derived from the data on SBMs collected in the participant diary.
Time Frame: Up to 24 hours after the first dose of study medication
Population: FAS included all participants randomized to receive study treatment whether or not they received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
percentage of participants | 60.0 | 41.5
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel — The proportion of participants with an SBM within 24 hours after first dose in Week 1 is analyzed by a Cochran-Mantel-Haenszel (CMH) test stratified by center. Centers with less participants were pooled based on geographical proximity; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.19 to 3.62]

4. Secondary Outcome: Mean Degree of Straining Score
Description: For each participant, the mean degree of straining was averaged for all SBMs in a given week. The degree of straining for each SBM was collected in the participant diary. The degree of straining was scored on a 5-point scale where: 0=No straining, 1=Mild straining, 2=Moderate straining, 3=Strong straining or 4=Very strong straining with higher scores indicating more severe straining.
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
score on a scale
  Week 1 | 1.6 (0.85) | 2.0 (0.88)
  Week 2 | 1.5 (0.89) | 1.8 (0.93)
  Week 3 | 1.3 (0.82) | 1.6 (0.92)
  Week 4 | 1.2 (0.92) | 1.5 (0.86)
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Week 1; Test type: Superiority; p = 0.001, Van Elteren Test — Average Degree of Straining was analyzed using Van Elteren Test stratified by center. Centers with less participants were pooled based on geographical proximity; Median Value of CI = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 2: Comparison: Lubiprostone 24 μg vs Placebo; Week 2; Test type: Superiority; p = 0.004, Van Elteren Test — [p-value comment as in outcome 4, analysis 1]; Median Value of CI = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 3: Comparison: Lubiprostone 24 μg vs Placebo; Week 3; Test type: Superiority; p = 0.024, Van Elteren Test — [p-value comment as in outcome 4, analysis 1]; Median Value of CI = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 4: Comparison: Lubiprostone 24 μg vs Placebo; Week 4; Test type: Superiority; p = 0.010, Van Elteren Test — [p-value comment as in outcome 4, analysis 1]; Median Value of CI = -0.3, 95% CI 2-sided [-0.5 to -0.1]

5. Secondary Outcome: Mean Degree of Stool Consistency
Description: For each participant, the mean stool consistency score was averaged for all SBMs in a given week. The mean degree of stool consistency for each SBM was collected in the participant diary based on the Bristol Stool Chart. The Bristol Stool Chart is a medical aid designed to classify the form of human feces into seven categories where: 1=Hard and round (difficult-to-pass), 2=Sausage-shaped but hard stool, 3=Sausage-shaped stool with cracks on the surface, 4=Sausage-shaped, soft stool with smooth surface, or coiled stool, 5=Soft, half-solid (and easy-to-pass) stool with clear crease, 6=Unshaped, loose stool with small, irregular-shaped pieces, or mushy stool or 7=Watery stool without solid pieces (entirely liquid).
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
score on a scale
  Week 1 | 4.1 (1.30) | 3.4 (1.08)
  Week 2 | 4.1 (1.13) | 3.5 (1.05)
  Week 3 | 4.1 (1.12) | 3.5 (0.93)
  Week 4 | 4.1 (1.19) | 3.6 (0.93)
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Week 1; Test type: Superiority; p < 0.001, Van Elteren Test — Mean Degree of Stool Consistency was analyzed using Van Elteren Test stratified by center. Centers with less participants were pooled based on geographical proximity; Median Value of CI = 0.6, 95% CI 2-sided [0.4 to 1.0]
Statistical Analysis 2: Comparison: Lubiprostone 24 μg vs Placebo; Week 2; Test type: Superiority; p < 0.001, Van Elteren Test — [p-value comment as in outcome 5, analysis 1]; Median Value of CI = 0.6, 95% CI 2-sided [0.4 to 0.9]
Statistical Analysis 3: Comparison: Lubiprostone 24 μg vs Placebo; Week 3; Test type: Superiority; p < 0.001, Van Elteren Test — [p-value comment as in outcome 5, analysis 1]; Median Value of CI = 0.6, 95% CI 2-sided [0.4 to 0.8]
Statistical Analysis 4: Comparison: Lubiprostone 24 μg vs Placebo; Week 4; Test type: Superiority; p < 0.001, Van Elteren Test — [p-value comment as in outcome 5, analysis 1]; Median Value of CI = 0.5, 95% CI 2-sided [0.2 to 0.7]

6. Secondary Outcome: Weekly Abdominal Symptoms Score
Description: Weekly abdominal symptoms of bloating and discomfort upon waking in the morning was scored weekly on a 5-point scale where: 0=None, 1=Mild, 2=Moderate, 3=Severe or 4=Very severe, with a higher score indicating more severe symptoms. Assessment of weekly abdominal symptoms were recorded in the participant in the diary.
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubiprostone 24 μg | Placebo
Number analyzed (Participants) | 105 | 106
score on a scale
  Week 1 | 1.4 (1.05) | 1.8 (0.96)
  Week 2 | 1.2 (0.93) | 1.5 (1.01)
  Week 3 | 1.0 (1.01) | 1.4 (0.93)
  Week 4 | 0.9 (0.94) | 1.2 (0.98)
Statistical Analysis 1: Comparison: Lubiprostone 24 μg vs Placebo; Week 1; Test type: Superiority; p = 0.020, Van Elteren Test — Abdominal Bloating was analyzed using Van Elteren Test stratified by center. Centers with less participants were pooled based on geographical proximity; Median Value of CI = -0.5, 95% CI 2-sided [-0.9 to -0.1]
Statistical Analysis 2: Comparison: Lubiprostone 24 μg vs Placebo; Week 2; Test type: Superiority; p = 0.072, Van Elteren Test — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Lubiprostone 24 μg vs Placebo; Week 3; Test type: Superiority; p < 0.001, Van Elteren Test — [p-value comment as in outcome 6, analysis 1]; Median Value of CI = -0.5, 95% CI 2-sided [-0.9 to -0.1]
Statistical Analysis 4: Comparison: Lubiprostone 24 μg vs Placebo; Week 4; Test type: Superiority; p = 0.004, Van Elteren Test — [p-value comment as in outcome 6, analysis 1]; Median Value of CI = -0.5, 95% CI 2-sided [-0.9 to -0.1]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to Week 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Lubiprostone 24 μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/106
Other Adverse Events (participants affected / at risk) | 23/105 | 19/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone 24 μg (N=105) | Placebo (N=106)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Influenza (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 4
Bronchitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT02729909/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT02729909/SAP_001.pdf